CLINICAL TRIAL: NCT03770780
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED CROSSOVER STUDY OF SAGE-718 USING A KETAMINE CHALLENGE, TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMIC RESPONSE USING MAGNETIC RESONANCE IMAGING IN HEALTHY SUBJECTS
Brief Title: A Study to Assess the Electrophysiology, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Response Using Magnetic Resonance Imaging of SAGE-718 Using a Ketamine Challenge in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 718-EXM-102
Record Dates: First submitted 2018-11-07; First posted 2018-12-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAGE-718 (Experimental)
  Interventions: Drug: SAGE-718
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718 in combination with Ketamine
  Arms: SAGE-718
Drug: Placebo — Placebo in combination with Ketamine
  Arms: Placebo

SUMMARY:
This study is a phase 1, double-blind, placebo-controlled crossover study of SAGE-718 using a ketamine challenge, to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic response using magnetic resonance imaging in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide 2 forms of identification; at least 1 must have a photo.
2. Subject has a body weight ≥50 kg and body mass index ≥18.0 and ≤30.0 kg/m2 at screening.
3. Subject is healthy with no history or evidence of clinically relevant medical disorders as determined by the Investigator.

Exclusion Criteria:

1. Subject has a history or presence of any psychiatric disease or condition including suicidal ideation or behavior, has answered YES to any question on the C-SSRS at screening or admission, or is currently at risk of suicide in the opinion of the Investigator
2. Subject has a history or presence of a neurologic disease or condition, including but not limited to epilepsy, closed head trauma with clinically significant sequelae, or a prior seizure.
3. Subject has a family history of epilepsy.
4. Subject has evidence of any metal in the body that may be contraindicated for receiving an MRI. This includes, but is not limited to: cardiac pacemaker, surgical implants, previous accident resulting in metal or shrapnel lodged internally, tattoos inked with metallic dyes, or a history of metal work without using protective eyewear.
5. Subject has claustrophobia or a history of claustrophobia.
6. Subject is unable or unwilling to remove piercings and/or jewelry that contain metal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Change in glutamate and glutamine (GLX) in the anterior cingulate cortex (ACC), hippocampus, and pons as measured with magnetic resonance spectroscopy (MRS) | Between Day 1 and Day 11

SECONDARY OUTCOMES:
Change in glutamate in the ACC, hippocampus, and pons, as measured with MRS | Between Day 1 and Day 11
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by incidence of adverse events (AEs)/serious AEs (SAEs) | Between Baseline and Day 27
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by electroencephalograms (EEGs) | Between Baseline and Day 27
  Observed values and change from baseline in EEGs in patients post study drug administration
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by electrocardiograms (ECGs) | Between Baseline and Day 27
  Observed values and change from baseline in ECGs in patients post study drug administration
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Between Baseline and Day 27
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by Brief Psychiatric Rating Scale (BPRS) | Between Baseline and Day 27
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by Clinician Administered Dissociative State Scale (CADSS) | Between Baseline and Day 27
Safety and tolerability of SAGE-718 alone and in combination with ketamine, as assessed by Observer's Assessment of Alertness and Sedation (OAAS) | Between Baseline and Day 27

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.